CLINICAL TRIAL: NCT01276197
Title: Using Stories to Address Disparities in Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 10-132
Record Dates: First submitted 2011-01-11; First posted 2011-01-13 (Estimated); Results first posted 2016-09-30 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-10

CONDITIONS: Hypertension
Keywords: hypertension; healthcare disparities; minority health; health behavior
MeSH Terms: conditions — Hypertension; Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Story-Telling DVD (Experimental): Participant will receive a DVD with informational and story-telling components
  Interventions: Other: Story-Telling DVD
- Arm 2: Non-Storytelling DVD (Active Comparator): Participant will receive an informational DVD
  Interventions: Other: Non-Storytelling DVD

INTERVENTIONS:
Other: Story-Telling DVD — DVD will contain both informational and story-telling components.
  Arms: Arm 1: Story-Telling DVD
Other: Non-Storytelling DVD — DVD will contain only informational component.
  Arms: Arm 2: Non-Storytelling DVD

SUMMARY:
The purpose of this study is to determine if patients with high blood pressure are better able to control their blood pressure after watching a DVD about blood pressure.

DETAILED DESCRIPTION:
This project consists of two phases: (1) Collecting of stories and creating a stories DVD; and (2) delivering the DVD in a randomized control trial (RCT). Both phases are described below.

The investigators will make two DVDs of African-American Veterans who will tell their success stories with controlling hypertension (HTN). The investigators want to help African-American Veterans control their hypertension by showing them stories that are interesting and that they can identify with, as well as giving them information about ways they can manage hypertension in their everyday lives. This is important because a disproportionate number of minority patients, including Veterans, have poorly controlled blood pressure. By showing them stories, rather than using more traditional methods of health education, the investigators hope to overcome some typical barriers to HTN control among the African-American population, including: lower levels of health literacy and numeracy, less trust in the medical system, and different (non-medical) models to explain their illness.

The Veteran storytellers will come from three VA sites (Charleston, Chicago, and Philadelphia) and their stories will be chosen based on (1) the proven effectiveness of the strategies they suggest for controlling BP and (2) how authentic they are, or how much they will "ring true" with the experiences of other Veterans, including their struggles and lessons learned.

After the DVD is complete, the investigators will conduct a randomized control trial to evaluate how effective it is in helping vets control their hypertension: 780 African-American vets with uncontrolled hypertension, from the same three VA sites, will participate. Half of them will watch the "Stories" DVD the investigators created; and the other half will watch a control, a DVD with the same medical information but without the narrative component. The investigators will measure their blood pressure (BP) just before they watch the DVD and again six months later. The investigators hypothesize that, six months after enrollment, the Veterans who watched the "Stories" DVD will have greater reduction in BP, as compared with those who watch the control. The investigators will also test the "Stories" DVD's impact on medication adherence and HTN management behaviors.

ELIGIBILITY:
Inclusion Criteria:

* African-American
* Diagnosis of HTN
* Uncontrolled BP as defined by BP >140/90 twice in the preceding 12 months

Exclusion Criteria:

* active substance abuse
* severe mental illness
* cognitive disabilities that might prevent them from actively or reliably participating in the interviews

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 618 (Actual)
Dates: Start 2013-01; Primary Completion 2015-05 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas K Houston, MD MPH, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA
Locations (4):
- United States (4):
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts
  - Philadelphia VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
We plan to report on our primary outcome

REFERENCES:
- [Result] Houston TK, Cherrington A, Coley HL, Robinson KM, Trobaugh JA, Williams JH, Foster PH, Ford DE, Gerber BS, Shewchuk RM, Allison JJ. The art and science of patient storytelling-harnessing narrative communication for behavioral interventions: the ACCE project. J Health Commun. 2011 Aug;16(7):686-97. doi: 10.1080/10810730.2011.551997. Epub 2011 May 24. PMID 21541875
- [Result] Fix GM, Bokhour BG. Understanding the context of patient experiences in order to explore adherence to secondary prevention guidelines after heart surgery. Chronic Illn. 2012 Dec;8(4):265-77. doi: 10.1177/1742395312441037. Epub 2012 Mar 2. PMID 22387691
- [Result] Fix GM, Houston TK, Barker AM, Wexler L, Cook N, Volkman JE, Bokhour BG. A novel process for integrating patient stories into patient education interventions: incorporating lessons from theater arts. Patient Educ Couns. 2012 Sep;88(3):455-9. doi: 10.1016/j.pec.2012.06.012. Epub 2012 Jul 6. PMID 22770814
- [Derived] Houston TK, Fix GM, Shimada SL, Long JA, Gordon HS, Pope C, Volkman J, Allison JJ, DeLaughter K, Orner M, Bokhour BG. African American Veterans Storytelling: A Multisite Randomized Trial to Improve Hypertension. Med Care. 2017 Sep;55 Suppl 9 Suppl 2:S50-S58. doi: 10.1097/MLR.0000000000000766. PMID 28806366

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Story-Telling DVD | Arm 2: Non-Storytelling DVD
Started | 308 | 310
Completed | 200 | 200
Not Completed | 108 | 110

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Story-Telling DVD | Arm 2: Non-Storytelling DVD | Total
Number analyzed (Participants) | 308 | 310 | 618
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 190 | 186 | 376
  >=65 years | 118 | 124 | 242
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 282 | 285 | 567
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 308 | 310 | 618
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Systolic BP at Follow-up
Description: Systolic Bp measurement at 6-month follow-up; we modeled the impact of Intervention assignment on SBP, adjusting for Baseline. Thus, baseline SBP was collected but not used as outcome; Baseline SBP us used as a covariate.
Time Frame: 6 months after intervention
Population: Our analyses was completed with those who completed follow-up visit and varies from participant flow as we are not able to include those lost to follow-up.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Arm 1: Story-Telling DVD | Arm 2: Non-Storytelling DVD
Number analyzed (Participants) | 264 | 270
mmHg | 137.9 (18.4) | 141.2 (17.8)

2. Primary Outcome: Diastolic BP Measurement at Follow-up
Description: Participants BP measurement at 6-month follow-up
Time Frame: 6-month following intervention
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Arm 1: Story-Telling DVD | Arm 2: Non-Storytelling DVD
Number analyzed (Participants) | 264 | 270
mmHg | 80.1 (13.0) | 81.9 (13.1)

ADVERSE EVENTS:
Arm/Group | Arm 1: Story-Telling DVD | Arm 2: Non-Storytelling DVD
Serious Adverse Events (participants affected / at risk) | 12/308 | 10/310
Other Adverse Events (participants affected / at risk) | 0/308 | 0/310
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Story-Telling DVD (N=308) | Arm 2: Non-Storytelling DVD (N=310)
Death (Congenital, familial and genetic disorders) | 2 (2) | 2 (2)
Hospitalization (Cardiac disorders) | 10 (10) | 8 (8)

LIMITATIONS AND CAVEATS:
Our multi-site trial was limited by challenges in recruitment (lower enrollment at one site) that resulted in overall recruitment lower than planned. Further, we did have some loss to follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes